CLINICAL TRIAL: NCT00978874
Title: [F18]EF5 PET/CT Imaging in Patients With Locally Advanced or Recurrent/Metastatic Carcinoma of the Cervix
Brief Title: Fluorine F 18 EF5 PET/CT Imaging in Patients With Locally Advanced or Recurrent/Metastatic Cervical Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is no longer with our institution
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 03808
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Fluorodeoxyglucose F18

ARMS (1):
- All subjects (Experimental)
  Interventions: Radiation: fludeoxyglucose F 18; Radiation: fluorine F 18 EF5

INTERVENTIONS:
Radiation: fludeoxyglucose F 18
Radiation: fluorine F 18 EF5

SUMMARY:
RATIONALE: Diagnostic procedures, such as fluorine F 18 EF5 PET/CT imaging, may help find oxygen in tumor cells. It may also help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This trial is studying fluorine F 18 EF5 PET/CT imaging to see how well it works in finding hypoxia in tumor cells of patients with locally advanced or recurrent/metastatic cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if the presence and heterogeneity of hypoxia can be detected by fluorine F 18 EF5 binding in tumors during PET/CT imaging in patients with newly diagnosed or recurrent carcinoma of the cervix.
* To determine if fludeoxyglucose F 18 uptake correlates with fluorine F 18 EF5 uptake.
* To assess the relationship between fluorine F 18 EF5 uptake and disease-free and overall survival.

OUTLINE: Patients are stratified according to disease stage (locally advanced vs recurrent or metastatic disease).

Patients receive fluorine F 18 EF5 IV followed by PET/CT imaging from the base of skull to upper thigh at baseline and during radiotherapy or chemotherapy (i.e., at 3-4 weeks after the initiation of radiotherapy or after the 4th, 5th, or 6th course of chemotherapy). Patients also undergo fludeoxyglucose F 18 PET/CT imaging within 7 to 10 days of the second fluorine F 18 EF5 scan.

After completion of study treatment, patients are followed up at 30 days and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of carcinoma of the cervix meeting 1 of the following criteria:

  * Pathologically confirmed, newly diagnosed stage IB-IVA (locally advanced) disease
  * Imaging evidence of recurrent or metastatic disease
* Measurable disease, defined as ≥ 1 cm on anatomic imaging

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* WBC > 2,000/mm³
* Platelet count > 90,000/mm³
* Total bilirubin < 2.0 mg/dL
* Creatinine < 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to Flagyl (metronidazole)
* No other condition or personal circumstance that, in the judgment of the Investigator, may interfere with the collection of complete, good-quality data

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2013-09-04 (Actual); Study Completion 2013-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilie Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: fludeoxyglucose F 18
  fluorine F 18 EF5
Period: Overall Study
Arm/Group | All Subjects
Started | 0 (The study was terminated and no data are available to be reported)
Completed | 0 (The study was terminated and no data are available to be reported)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and despite all possible attempts to contact the PI/study team, no data are available to be reported
Arm/Group | All Subjects
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Fluorine F 18 EF5 Uptake and Disease-free Survival and Overall Survival
Description: The study was terminated and no data are available to be reported
Time Frame: 7 years
Population: The study was terminated and no data are available to be reported
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: The study was terminated and no data are available to be reported
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes